CLINICAL TRIAL: NCT03949712
Title: Effects of Transcranial Static Magnetic Field Stimulation (tSMS) on Motor Learning and Cortical Neurophysiology in the Developing Brain
Brief Title: Pediatric Transcranial Static Magnetic Field Stimulation to Improve Motor Learning
Acronym: PSTIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Adam Kirton, Professor of Pediatrics, Radiology, and Clinical Neurosciences; Director of Calgary Pediatric Stroke Program and N3; Pediatric Neurologist, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: REB18-0178
Record Dates: First submitted 2019-04-18; First posted 2019-05-14 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Healthy; Pediatrics

STUDY DESIGN:
Intervention Model Description: Participants will receive all 3 treatment arms (Right M1 tSMS, Left M1 tSMS, sham tSMS) in a randomized order.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right motor cortex (M1) tSMS (Experimental): tSMS will be applied to the right motor cortex for 30 minutes.
  Interventions: Device: Transcranial Static Magnetic Field Stimulation (tSMS)
- Left motor cortex (M1) tSMS (Experimental): tSMS will be applied to the left motor cortex for 30 minutes.
  Interventions: Device: Transcranial Static Magnetic Field Stimulation (tSMS)
- Sham tSMS (Sham Comparator): Sham tSMS will be applied to the left or right motor cortex (randomized) for 30 minutes.
  Interventions: Device: Sham Transcranial Static Magnetic Field Stimulation (tSMS)

INTERVENTIONS:
Device: Transcranial Static Magnetic Field Stimulation (tSMS) — tSMS consists of a small compact cylindrical neodynium magnet (S-45-30-N, Supermagnete) with an estimated strength of up to 0.5 Tesla and a size of 30 mm x 45 mm.
  Arms: Left motor cortex (M1) tSMS; Right motor cortex (M1) tSMS
Device: Sham Transcranial Static Magnetic Field Stimulation (tSMS) — Sham tSMS consists of a small compact metal cylinder, identical in appearance to the real tSMS device.
  Arms: Sham tSMS

SUMMARY:
Non-invasive brain stimulation (NIBS) is a safe, painless way to improve brain function. It is used for many conditions, including to help children with disabilities. However, it can be challenging to apply NIBS in very young children and infants. A new, simple form of NIBS called transcranial static magnetic field stimulation (tSMS) is a promising tool for early brain stimulation. tSMS in adults has been shown to be safe, tolerable and have the desired effects on brain activity when applied to the motor cortex of the brain. However, how tSMS affects on motor function is not understood. This research will use tSMS to target the motor cortex which is responsible for voluntary movement. The study will determine if tSMS can improve motor learning in healthy children. It is hypothesized that application of tSMS on the right motor cortex will decrease excitability of the motor cortex and will lead to improved motor learning in the right hand. tSMS has the potential to become a safe, inexpensive, home-based way to enhance personalized rehabilitation for disabled children.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent/assent
2. age between 8 and 18 years
3. right-handedness
4. normal development
5. absence of neuropsychiatric diagnoses or medications

Exclusion Criteria:

1. diagnosis of a neurological, psychiatric or developmental disorder
2. metal in mouth, implanted pacemakers, or other contraindications for brain stimulation
3. confirmed or potential pregnancy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in amplitude of motor evoked potentials (MEPs) | Change from baseline to immediately following the tSMS intervention
  Baseline data will be collected through application of single Transcranial Magnetic Stimulation (TMS) pulses used to assess cortical excitability within one hemisphere. For this, two stimulators (Magstim and Bistim) are connected by an adaptor. A single flat iron Magnstim TMS coil is held over the right hotspot, and pairs of pulses is delivered from this coil. 10 test pulses at an intensity of 120% of resting motor threshold (RMT) are applied. These pulses will be randomized with other paired-pulses to collect other outcome measures (described in the secondary outcome measures section)

SECONDARY OUTCOMES:
Change in left-hand Purdue Pegboard Test (PPT) score. | Change in left-hand Purdue Pegboard Test (PPT) score from baseline to after the tSMS intervention
  A "baseline" trial will be performed. During the intervention, participants will perform 25 repetitions. A "post" trail will be performed following the neurophysiology measurements after the tSMS intervention. An increase in score on the PPT would be indicative of improved performance on the task.
Change in short-interval intracortical inhibition (SICI) | Change from baseline to immediately following the tSMS intervention
  Baseline data will be collected through application of paired TMS pulses used to assess cortical excitability within one hemisphere. For this, two stimulators (Magstim and Bistim) are connected by an adaptor. A single flat iron Magnstim TMS coil is held over the right hotspot, and pairs of pulses is delivered from this coil. A conditioning pulse is applied to the left hemisphere at an intensity of 80% RMT, followed by a test pulse over the right hemisphere at an intensity of 120% RMT. 10 pairs of pulses are applied with an interstimulus interval of 2 ms to test for SICI These pulses will be randomized with other paired-pulses and single pulses to collect other outcome measures (described in the primary and secondary outcome measures section)
Change in intracortical facilitation (ICF) | Change from baseline to immediately following the tSMS intervention
  Baseline data will be collected through application of paired TMS pulses used to assess cortical excitability within one hemisphere. For this, two stimulators (Magstim and Bistim) are connected by an adaptor. A single flat iron Magnstim TMS coil is held over the right hotspot, and pairs of pulses is delivered from this coil. A conditioning pulse is applied to the left hemisphere at an intensity of 80% RMT, followed by a test pulse over the right hemisphere at an intensity of 120% RMT. 10 pairs of pulses are applied with an interstimulus interval of 10 ms to test for ICF. These pulses will be randomized with other paired-pulses and single pulses to collect other outcome measures (described in the primary and secondary outcome measures section)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kirton, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Oliviero A, Mordillo-Mateos L, Arias P, Panyavin I, Foffani G, Aguilar J. Transcranial static magnetic field stimulation of the human motor cortex. J Physiol. 2011 Oct 15;589(Pt 20):4949-58. doi: 10.1113/jphysiol.2011.211953. Epub 2011 Aug 1. PMID 21807616
- [Background] Oliviero A, Carrasco-Lopez MC, Campolo M, Perez-Borrego YA, Soto-Leon V, Gonzalez-Rosa JJ, Higuero AM, Strange BA, Abad-Rodriguez J, Foffani G. Safety Study of Transcranial Static Magnetic Field Stimulation (tSMS) of the Human Cortex. Brain Stimul. 2015 May-Jun;8(3):481-5. doi: 10.1016/j.brs.2014.12.002. Epub 2014 Dec 11. PMID 25595064